CLINICAL TRIAL: NCT03859583
Title: Capsaicin Consumption on Resting Energy Expenditure and Glucose Metabolism
Brief Title: Capsaicin Energy Expenditure and Glucose Metabolism
Acronym: CAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, lilian de Jonge, assistant professor, George Mason University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1157054-1
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: capsaicin; resting metabolic rate; glucose
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsaicin (Experimental): 4 tsp of cayenne pepper in a 60g omelette
  Interventions: Dietary Supplement: Capsaicin
- Control (Placebo Comparator): 60 g omelette
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Capsaicin — 4 tsp of cayenne in a breakfast omelette
  Arms: Capsaicin
Dietary Supplement: Control — breakfast omelette without cayenne pepper
  Arms: Control

SUMMARY:
The aim of the study is to investigate the effects of capsaicin rich foods on resting energy expenditure and substrate oxidation. We plan to recruit 30 healthy lean and overweight individuals age 18-45 (women) and age 18-50 (men) who will undergo two test days in random order. During one day they will receive a breakfast of toast, orange juice and an omelette with 4tsp of cayenne pepper while on the other day they will receive the same breakfast without the cayenne pepper. Metabolic rate and Respiratory quotients is measured for 30 minutes before the meal and for 2 hours after the meal. Capillary glucose levels and heart rate and blood pressure are measured before the meal and every 30 minutes thereafter for 2 hours.

DETAILED DESCRIPTION:
Participants will be recruited by posters distributed on campus bulletin boards and asked to contact the investigator by phone or e-mail. Participants will complete a screening questionnaire by phone to determine eligibility. Once they pass the screening, they will be invited to the laboratory to sign the consent form, which will be administered by Rafia Virk. They will also be given a demographic survey. The survey will inquire about height, weight, medical conditions, medications and inclusion/exclusion criteria and availability. This survey will be used for screening purposes only and will not contribute to the research data. The survey is included in this application and inclusion and exclusion criteria are outlined. If participants are determined eligible, they will be contacted to set up with two study visits, pre-test instructions will be provided.

*For both appointments, participants will arrive to the test location after a 12-hour fast.

Appointment 1: Participants will arrive at the Nutrition Assessment Laboratory between 7:00am and 7:30am. Details of the study will be re-iterated and informed consent will be obtained first thing on the morning of the first appointment. Eligibility will then then be confirmed by measuring height and weight and BMI calculation, and a over the counter pregnancy test will be performed on women. Demographic survey and 24-hour dietary recall will be obtained for 2 week days and 1 weekend day. Baseline measurements will then be obtained which include: Waist circumference, body compositition by Dual Energy X-ray Absorptiometry (DXA) scan (performed by Dr. de Jonge or Rafia Virk, who will be trained by Dr. de Jonge). The DXA scan involves lying on a table while wearing lose fitting, comfortable clothing. The scanner uses a low dose x-ray to determine the amount of fat, muscle and bone in your body. After lying down for 30 minutes, a metabolic cart will be used to measure resting energy expenditure by indirect calorimetry. For this procedure, a plastic dome will placed over the participants head that will measure their resting energy expenditure (REE). Baseline REE will then be measured for 30 minutes. After getting a baseline measure participants will consume a standard meal. We will continue to measure resting energy expenditure for 120 minutes. Blood glucose using a glucometer will also be determine before and 2 hours after the standardized meal. The REE measurements will be performed by Ms. Rafia Virk. Ms. Virk will be trained in the use of the metabolic cart by Dr. Lilian de Jonge who has over 20 years experience in the use of indirect calorimetry for the assessment of REE. After this test, the subjects will undergo a capsaicin threshold test. For this test, deionized water with red food coloring will serve as the blank. The testing compound will be cayenne pepper. The target samples, containing very low concentrations of cayenne pepper (0-1mg/g), will also have red food coloring so that they will only be distinguishable to participant by sense of taste rather than taste and sight. There will be nine sets of rows, each with 3 sets of samples. Each set will contain 2 blanks and one target sample. The target sample increase in concentration as the participant moves along the row. The participant will be asked to taste test the samples and pick the target sample out of the three. This appointment will take about 3 hours.

The second test day will occur within one week of the first day. The participant will arrive with a 12 hour fast during the first week of the study. They will consume the same standardized meal (provided by Dr. de Jonge) from first appointment but with the addition of capsaicin (cayenne pepper powder form) (4tsp). They will then undergo a metabolic cart test (120 mins). Their blood glucose will also be determined using a glucometer for the following 3 hours post consumption. This appointment will last about 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age females or 18-50 males

  * Generally healthy non-diabetic overweight or obese men and women
  * BMI 23-33 kg/m2
  * Willing to abstain from caffeine and alcohol for 3 days prior to testing
  * Able to provide written consent in English
  * Ability to communicate in English (oral and written)

Exclusion Criteria:

* BMI < 23 kg/m2 or >33 kg/m2

  * Pregnant or Nursing
  * Taking prescribed or over the counter medication affecting fluid balance or metabolism
  * Suffers from hepatic, renal, pulmonary, endocrine or hematological disease
  * Performs more than 3 hours a week of strenuous exercise
  * Consumes, on average, more than 2 alcoholic beverages per day
  * More than 5 kg of weight change over the past 6 months
  * Claustrophobic
  * Consumes capsaicin foods habitually 3x/week

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Postprandial substrate oxidation | 3 hours
  The change in substrate oxidation after a meal as measured by the ratio of carbondioxide production and oxygen consumption measured by indirect calorimetry

SECONDARY OUTCOMES:
postprandial energy expenditure | 3 hrs
  Change in resting energy expenditure after meal consumption as measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided